CLINICAL TRIAL: NCT05619848
Title: Effect of Paravertebral Muscle Fat Infiltration on Rocuronium Use in Lumbar Surgery
Acronym: RUILS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zheng Guo (Other)
Responsible Party: Sponsor-Investigator, Zheng Guo, Ph.D., Second Hospital of Shanxi Medical University
Organization: Second Hospital of Shanxi Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: yuewei20221109
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Spinal Stenosis Lumbar
MeSH Terms: interventions — Rocuronium; Midazolam; Propofol; Etomidate; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild fat infiltration (Experimental): Fat infiltration rate is less than 30%
  Interventions: Drug: Rocuronium Bromide
- Moderate fat infiltration (Experimental): Fat infiltration rate is 30%~50%
  Interventions: Drug: Rocuronium Bromide
- Server fat infiltration (Experimental): Fat infiltration rate is greater than 50%
  Interventions: Drug: Rocuronium Bromide

INTERVENTIONS:
Drug: Rocuronium Bromide — 0.6 mg/kg rocuronium was injected intravenously, and rocuronium was pumped during operation to maintain deep muscle relaxation
  Other Names: Midazolam, propofol, etomidate and remifentanil

SUMMARY:
To investigate the effect of different degrees of fat infiltration on rocuronium use in lumbar surgery was monitored by trapezius muscle relaxation.

DETAILED DESCRIPTION:
Select the patients who will receive posterior lumbar surgery in the Second Hospital of Shanxi Medical University. According to the classification criteria of fat infiltration, it will be divided into three groups: mild, moderate and severe. This study will pump and titrate rocuronium bromide under the monitoring of muscle relaxation during the operation, record the dosage of rocuronium bromide and the duration of pump injection, and evaluate its clinical effect. Postoperative results include the use and clinical effect of rocuronium, which will be counted after the trial.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-65; ASA grade I-II; no significant cardiopulmonary disease; no history of surgery in the corresponding surgical area; no coagulopathy.

Exclusion Criteria:

refusal to participate by the present experimenter; those with severe cardio-cerebrovascular disease, severe hepatic and renal dysfunction; taking medications affecting the neuromuscular junction; area of monitoring site for skin breakers; patients with intraoperative bleeding, anaphylactic shock, or other serious complications; patients requiring intraoperative neurophysiological monitoring (including sensory, motor evoked potentials).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
use of rocuronium bromide | Perioperative period
  average dosage

SECONDARY OUTCOMES:
The general condition of the paraspinal muscle | Perioperative period
  Fat infiltration rate

OTHER OUTCOMES:
Muscle relaxation satisfaction score | Perioperative period
  satisfaction score

CONTACTS AND LOCATIONS:
Overall Officials: Guo Zheng, Ph. D, Study Chair — Second of Shanxi Medical University
Locations (1):
- Second of Shanxi Medical University, Taiyuan, Shanxi, China